CLINICAL TRIAL: NCT04608448
Title: An Innovative Proof-of-concept Approach to Identify Age-modulating Drugs Capable of Reversing Inflammation and Re-setting the Epigenetic Clock (Topical-RAPA)
Brief Title: Topical-RAPA Use in Inflammation Reversal and Re-setting the Epigenetic Clock
Acronym: Topical-RAPA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ellen Kraig, Prof & Deputy Chair of Faculty Development Cell Systems & Anatomy, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20200720H; 1R21AG068731-01 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Aging; Epigenetics; Inflammatory Mediators
Keywords: Epigenetic clock
MeSH Terms: interventions — Petrolatum

STUDY DESIGN:
Intervention Model Description: Participants will be their own control, either right or left arm will be randomized to treatment or placebo.
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed by the compounding pharmacy. Ointment dispensers will be color-coded for left and right arm for each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Rapamycin (Active Comparator): Ointment is applied to a color coded area on the subject forearm daily.
  Interventions: Drug: Rapamycin Topical Ointment
- Placebo (Placebo Comparator): Placebo ointment is applied to a color coded area on the subject forearm daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rapamycin Topical Ointment — 8% topical rapamycin ointment
  Other Names: Sirolimus Topical Ointment; RAPA Topical Ointment
  Arms: Topical Rapamycin
Other: Placebo — Petrolatum ointment containing no active ingredient
  Other Names: Placebo Topical Ointment; Petrolatum
  Arms: Placebo

SUMMARY:
Topical Rapamycin ointment will be applied to participant forearms to test whether epigenetic changes in the skin are elicited.

DETAILED DESCRIPTION:
Rapamycin 8% ointment will be applied topically to one of the participant's forearms and matching placebo to the opposite forearm daily for a total of 6 months. After consenting, screening and randomization of arms, the participants will be monitored at monthly visits until study completion.

ELIGIBILITY:
Inclusion Criteria:

* 65-95 years of age.
* Good health with all chronic diseases (hypertension, coronary artery disease, etc.) clinically stable.
* Selected subjects will be in good health (Per the World Health Organization, good health will be defined as complete physical, mental, and social well-being and not merely the absence of disease or infirmity).
* All diseases or infirmities will be clinically stable whether managed by medications or not.
* CLOX score of 10 or greater
* Women will be postmenopausal
* Postmenopausal women taking hormone replacement will be included if they have been on a stable dose for ≥6 months
* Live within a 20 mile drive of the UTHSA campus (7703 Floyd Curl Drive, San Antonio, TX)

Exclusion Criteria:

* Diabetes.
* History of skin ulcers or poor wound healing, or keloid formers.
* Smoking.
* Liver disease.
* Coumadin anti-coagulation.
* Treatment with drugs known to affect cytochrome P450 3A (diltiazem, erythromycin, etc. - due to role in rapamycin metabolism).
* Treatment with an immunosuppressant (prednisone, etc.) within 6 months.
* History of recent (within 6 months) Myocardial Infarction or active Coronary Disease.
* Hypersensitivity to rapamycin or petrolatum (ointment vehicle)
* Arm tattoos or scars in application area

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kraig, PhD, Principal Investigator — University of Texas Health at San Antonio; Dean L Kellogg, Jr., MD, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Unidentified IPD will be shared in publication form in peer-reviewed journals, at national or international meetings and with collaborating investigators at the PIs home institution.
  Summary results will be published on ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared upon study completion.
Access Criteria: Will be provided upon formal request to PI and/or included in publications.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects acted as their own controls, one forearm had rapamycin ointment applied and the other placebo, thus there were 20 participants who had both rapamycin applied to one arm and placebo to the other.
Units Other Than Participants: Forearms of subjects
Groups:
- Topical Rapamycin Applied to One Arm and Placebo Applied to the Opposite Arm: Ointment is applied to a color coded area on the subject forearm daily.
  Rapamycin Topical Ointment: 8% topical rapamycin ointment
Period: Overall Study
Arm/Group | Topical Rapamycin Applied to One Arm and Placebo Applied to the Opposite Arm
Started | 22; 44 Forearms of subjects
Completed | 20; 40 Forearms of subjects
Not Completed | 2; 4 Forearms of subjects
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Each subject applied either an ointment containing the mTOR inhibitor rapamycin or a vehicle-only control ointment to a 1 cm patch of skin on the forearm daily for 6 months and a placebo applied to the opposite arm.
Groups:
- Topical Rapamycin: Ointment is applied to a color coded area on the subject forearm daily.
  Rapamycin Topical Ointment: 8% topical rapamycin ointment to one arm and Petrolatum ointment containing no active ingredient to the opposite arm
Arm/Group | Topical Rapamycin
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants] — Population: Each subject applied either an ointment containing the mTOR inhibitor rapamycin or a vehicle-only control ointment to a 1 cm patch of skin on the forearm daily for 6 months.
  Participants
    Age 65-92 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Epigenetic Markers
Description: A set of DNA methylation marks that correlate with chronological age will be used to measure rejuvenation of the "epigenetic clock" due to drug treatment compared to placebo. Using Illumina EPIC arrays, CpG methylation will be assessed and then the predicted age, based on the combined methylation at the set of 391 marks (the "epigenetic clock" as defined by Dr. Steven Horvath, UCLA), will be determined.
Time Frame: Baseline to 6 months
Population: DNA prepared from the placebo and rapamycin-treated skin sites was analyzed for methylation at specific sites known to change with age.
Measure: Mean (Full Range); unit: years
Units Other Than Participants: Forearm of participant
Arm/Group | Topical Rapamycin | Placebo
Number analyzed (Participants) | 20 | 20
Number analyzed (Forearm of participant) | 20 | 20
years | 84.4 [66.2 to 109.8] | 82.8 [64.3 to 98.1]

2. Secondary Outcome: Change in Inflammatory Marker IL-6
Description: A measure of inflammatory markers will include analytes that are affected either by aging or oral rapamycin. Inflammatory markers are measured using Enzyme-Linked Immuno-Sorbant Assays (ELISA). The marker to be measured is IL-6.
Time Frame: Baseline to 6 months
Population: Recovery of blister fluid from some subjects was lower than anticipated so a Luminex-based array assay, which uses much lower sample volumes than ELISAs, was performed and the cytokine levels on the rapamycin treated side were compared to the placebo levels.
Measure: Mean (Full Range); unit: pg/ml
Units Other Than Participants: Blisters
Arm/Group | Topical Rapamycin | Placebo
Number analyzed (Participants) | 16 | 16
Number analyzed (Blisters) | 16 | 16
pg/ml | 1.44 [0 to 11.74] | 1.57 [0 to 7.97]

3. Secondary Outcome: Change in Inflammatory Marker CRP
Description: A measure of inflammatory markers will include analytes that are affected either by aging or oral rapamycin. Inflammatory markers are measured using Enzyme-Linked Immuno-Sorbant Assays (ELISA). The marker to be measured is CRP. No data were obtained from this measure due to the low blister fluid volume.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to 6 months
Description: Adverse events are reported per subject arm, since each subject had both rapamycin applied to one arm and placebo to the other arm
Groups:
- Placebo: Placebo ointment is applied to a color coded area on the subjects' opposite forearm daily.
Arm/Group | Topical Rapamycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Rapamycin (N=22) | Placebo (N=22)
Rash/redness (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) — Rash at site of application

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04608448/Prot_SAP_002.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT04608448/ICF_001.pdf